CLINICAL TRIAL: NCT05455463
Title: Effect of Participation in Virtual Exercise Sessions on Physical Activity, Language and Cognitive Functioning, and Quality of Life in Persons With Aphasia
Brief Title: Effect of Participation in Virtual Exercise Sessions in Persons With Aphasia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: California State University, East Bay (Other)
Responsible Party: Principal Investigator, Michelle Gravier, Assistant Professor, California State University, East Bay
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: CSUEB-IRB-2020-83
Record Dates: First submitted 2022-06-30; First posted 2022-07-13 (Actual); Last update posted 2024-02-06 (Actual); Status verified 2024-02

CONDITIONS: Aphasia, Acquired
MeSH Terms: conditions — Aphasia

STUDY DESIGN:
Intervention Model Description: Participants who elect to take part in the exercise intervention will be assigned to the intervention group, while those who do not will be assigned to the control group.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Online aphasia-adapted physical activity class (Experimental): Will receive the physical activity intervention.
  Interventions: Behavioral: Online aphasia-adapted physical activity class
- Usual routine control (No Intervention): Engage in physical activity per usual routine.

INTERVENTIONS:
Behavioral: Online aphasia-adapted physical activity class — Online 50-minute physical activity sessions, two to three times weekly for 10-11 weeks. The activity instructions will be modified to be aphasia-friendly (simplified language, multimodality support).
  Arms: Online aphasia-adapted physical activity class

SUMMARY:
The purpose of this study is to test the feasibility and acceptability of an online exercise program for community-dwelling individuals with aphasia, a language disorder resulting from brain damage. Physical activity, language, cognitive, and quality of life outcomes will be collected to assess potential effectiveness.

DETAILED DESCRIPTION:
Approximately one-third of stroke survivors have aphasia, acquired language difficulty that affects the ability speak and understand others. However, despite documented benefits of interventions to promote physical activity (PA) after stroke, including improved health-related quality of life (QoL), social and emotional benefits, and improved cognition, individuals with aphasia are often excluded from this research due to their communication difficulties. This is particularly concerning, given that individuals with aphasia are at greater risk of social isolation and depression compared to stroke survivors without aphasia. Presently, limited research has been conducted that examines the effect of PA interventions in individuals with aphasia although preliminary findings suggest that benefits may exist across domains (health and disability).

This study aims to better understand how PA affects the lives of individuals with aphasia. Given weekly tele-instruction in PA over 10 weeks, participants' levels of PA will be monitored for the duration of the study. Pre- and post-treatment measures of cognitive ability, QoL, and aphasia severity will be collected and analyzed to characterize intervention effects. The results of this study will provide insight into whether PA may be an important component of future aphasia treatment.

ELIGIBILITY:
Inclusion Criteria:

* Presence of aphasia
* Able to join exercise classes over Zoom

Exclusion Criteria:

* None

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 28 (Actual)
Dates: Start 2020-09-17 (Actual); Primary Completion 2023-12-31 (Actual); Study Completion 2023-12-31 (Actual)

PRIMARY OUTCOMES:
Adherence Rates | During intervention (weeks 1-10)
  Percent of classes attended
Retention | Post-intervention (week 10)
  Percent of participants completing the intervention

SECONDARY OUTCOMES:
Participants' attitudes towards the intervention | Post-intervention (week 10)
  Acceptability and themes as identified via qualitative interview

OTHER OUTCOMES:
Sedentary behaviors | Pre-intervention (week 0) and post intervention (week 10)
  Change in sitting and sleeping time, as measured using activity monitor
Physical Activity: Steps | Pre-intervention (week 0) and post intervention (week 10)
  Change in steps per day, as measured using activity monitor
Physical Activity: Standing | Pre-intervention (week 0) and post intervention (week 10)
  Change in time spent standing, as measured using activity monitor
Engagement | During intervention (weeks 1-10)
  Change in heart rate during exercise class, as measured using activity monitor
Language ability | Pre-intervention (week 0) and post intervention (week 10)
  Change in Western Aphasia Battery-Revised Aphasia Quotient (minimum value:0, maximum value: 100, higher scores indicate a better outcome)
Quality of Life (perceived) | Pre-intervention (week 0) and post intervention (week 10)
  Change in Burden of Stroke Scale Total Transformed Score; minimum value 0; maximum value 100; higher scores indicate worse outcome
Cognition | Pre-intervention (week 0) and post intervention (week 10)
  Change in Test of Non-Verbal Intelligence Percentile Rank (minimum score: 0, maximum score 100, higher scores indicate a better outcome)

CONTACTS AND LOCATIONS:
Overall Officials: Michelle 1 Gravier, Ph.D., Principal Investigator — California State University, East Bay
Locations (1):
- California State University, East Bay, Hayward, California, United States

IPD SHARING:
Plan to Share IPD: Yes
De-identified data will be made available upon reasonable request
Supporting Information: Study Protocol, ICF
Time Frame: Data will become available at study conclusion and will be available for 7 years.
Access Criteria: Requests received by the primary investigator or other investigator team members via email will be reviewed for reasonable use